CLINICAL TRIAL: NCT02160327
Title: The Role of Cytokines and Mast Cell in the Pathogenesis of Ocular Surface Inflammation Diseases Including Superior Limbic Keratoconjunctivitis, Conjunctivochalasis, and Dry Eye
Brief Title: The Role of Cytokines and Mast Cell in the Pathogenesis of SLK, Conjunctivochalasis, and Dry Eye
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201312127RINB
Record Dates: First submitted 2014-05-27; First posted 2014-06-10 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Superior Limbic Keratoconjunctivitis; Conjunctivochalasis; Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * tear
  * conjunctival tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
The specific aims of the the investigators studies are as follows:

* To collect the tear samples from patients with different ocular surface disorders, including SLK, conjunctivochalasis, and keratoconjunctivitis sicca (KCS).
* To evaluate the differential expression of tear cytokines and pH values between different ocular surface disorders.
* To collect the surgical conjunctival specimens from the patients with SLK and conjunctivochalasis.
* To evaluate the factors inducing mast cell migration and how mast cell is activated in SLK via surgical specimens and cultivated fibroblast.

DETAILED DESCRIPTION:
1. Detection of various tear cytokine levels in patients with superior limbic keratoconjunctivitis, conjunctivochalasis, and keratoconjunctivitis sicca

   - Basal tear samples will be collected atraumatically from the inferolateral tear meniscus by using glass capillary tubes. Care is taken to avoid touching the corneal and conjunctival surface. Approximately 30 μl of tear samples is obtained, and then the samples are centrifuged for 10 minutes at 1500 rpm (225g). Tear sample are placed in microtubes (Eppendorf) and stored at -70°C. IL-1β, IL-17, TNF-α, and IFN-γ levels will be measured by enzyme-linked immunosorbent assay kits.
2. Immunohistochemistry stain method for conjunctival specimens - The conjunctiva will be collected from SLK and conjunctivochalasis patients who received superior and inferior bulbar conjunctival resection as needed. The redundant conjunctiva noted after peritomy during cataract or retinal surgery will be excised to serve as a normal control. The conjunctival specimens of all the SLK, conjunctivochalasis, and control groups are sent to the pathology department for routine paraffin embedding and hematoxylin and eosin staining. The surgical specimens are placed into 4% paraformaldehyde at 4 C for one to two days and then stored in 1% sodium phosphate buffer at 4 C. They then are embedded in paraffin. To enhance tissue adhesion, 5-micrometer thick sections are mounted on glass slides pre- treated with Vectabond (Vector Laboratories, Burlingame, California, USA). The paraffin sections are deparaffinized, rehydrated and washed with phosphate-buffered saline (PBS; pH 7.4). Antigen retrieval is performed by immerse the sections in 0.1% trypsin in water bath for 15 mins. The endogenous peroxidase activity is quenched by placing the slides in 3% hydrogen peroxide. The slides are then blocked with serum followed by incubation with primary antibodies. Primary antibodies (TSL and SCF) are incubated overnight at 4°C. Thereafter, incubation with biotin conjugated secondary antibody is performed at room temperature for 60 min. Further, incubation with avidin-biotin horseradish peroxidase complex is then performed at room temperature as well for 30 min using Vectastain elite® ABC kit (Vector labs, CA USA). The location where the enzyme is bound will be visualized by the addition of the substrate 3,3'-diaminobenzidine (DAKO, CA, USA), a chromogen which produces a brown insoluble precipitate. The sections are then counterstained with haematoxylin, which is followed by dehydration and mounting with Vecta Mount Mounting medium was used to evaluate the slides.

ELIGIBILITY:
• Part I. Tear sample

Inclusion criteria:

1. age 20-85 years old
2. diagnosed as a patients of superior limbic keratoconjunctivitis (SLK) or conjunctivochalasis or keratoconjunctivitis sicca (KCS)

Exclusion criteria:

1. pregnancy
2. any ocular surgery within 3 months

   * Part II. Surgical conjunctiva specimen

Inclusion criteria:

1. age 20-85 years old
2. disease group: SLK or conjunctivochalasis patients refractory to medical treatment and receiving conjunctival resection surgery
3. control group: patients receiving retinal or cataract surgery with redundant conjunctiva after peritomy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part I. Tear sample diagnosed as a patients of superior limbic keratoconjunctivitis (SLK) or conjunctivochalasis or keratoconjunctivitis sicca (KCS) Part II. Surgical conjunctiva specimen disease group: SLK or conjunctivochalasis patients refractory to medical treatment and receiving conjunctival resection surgery
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Tear cytokines change measured by ELISA | Tear will be collected before treatment, one month and six months follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Fung-Rong Hu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan